CLINICAL TRIAL: NCT00473967
Title: Double-blind, Randomized, Controlled Phase 1 Study of the Safety and Immunogenicity of Na-ASP-2 Hookworm Vaccine in Previously-Infected Brazilian Adults
Brief Title: Phase 1 Trial of Na-ASP-2 Hookworm Vaccine in Previously Infected Brazilian Adults
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Occurrence of unacceptable adverse events.
Sponsor: Albert B. Sabin Vaccine Institute (Other)
Collaborators: Oswaldo Cruz Foundation (Other); George Washington University (Other); London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SVI-06-02
Record Dates: First submitted 2007-05-14; First posted 2007-05-16 (Estimated); Last update posted 2012-07-09 (Estimated); Status verified 2012-07

CONDITIONS: Hookworm Infection
Keywords: Vaccine; Hookworm; Phase 1; Na-ASP-2
MeSH Terms: conditions — Hookworm Infections; Ancylostomiasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 10 mcg Na-ASP-2/Alhydrogel (Experimental): Na-ASP-2 Hookworm Vaccine
  Interventions: Biological: Na-ASP-2 Hookworm Vaccine
- Butang hepatitis B vaccine (Active Comparator): Hepatitis B Vaccine - comparator vaccine
  Interventions: Biological: Na-ASP-2 Hookworm Vaccine

INTERVENTIONS:
Biological: Na-ASP-2 Hookworm Vaccine — Injections of one of three different dose concentrations of the Na-ASP-2 vaccine (10, 50, or 100 mcg) vs. the hepatitis B vaccine, delivered at 0, 2, and 4 months by intramuscular injection.

SUMMARY:
Na-ASP-2 is a protein expressed during the larval stage of the N. americanus hookworm life cycle. Vaccination with recombinant ASP-2 has protected dogs and hamsters from infection in challenge studies. In a clinical study in hookworm-uninfected adults in the USA, Na-ASP-2 Hookworm Vaccine was safe and immunogenic. This study will evaluate its safety and immunogenicity in individuals living in an area of endemic hookworm infection.

DETAILED DESCRIPTION:
* Double-blind, randomized, controlled Phase 1 clinical trial.
* Study site: Americaninhas, Minas Gerais, Brazil.
* Number of participants: 48 in three groups of 16, randomized to receive either Na-ASP-2 Hookworm Vaccine (n=36) or Butang® hepatitis B vaccine (n=12).
* Study duration: 48 weeks; each participant will be followed for a total of 42 weeks.
* Immunization schedule: Study days 0, 56 and 112.
* Route: IM in the deltoid muscle.
* Dose of Na-ASP-2: 10, 50 and 100 µg for the first, second and third dose cohort, respectively.
* Dose of Alhydrogel®: 800 µg for each dose of Na-ASP-2.

ELIGIBILITY:
Inclusion Criteria:

* Males or females between 18 and 45 years, inclusive.
* Known residents of the Municipality of Novo Oriente de Minas, Minas Gerais, Brazil.
* Good general health as determined by means of the screening procedure.
* Completed a 3-dose albendazole treatment for documented hookworm infection during the previous 3 months.
* Available for the duration of the trial (42 weeks).
* Willingness to participate in the study as evidenced by signing the informed consent document.

Exclusion Criteria:

* Pregnancy as determined by a positive urine β-hCG (if female).
* Participant unwilling to use reliable contraception methods up until one month following the third immunization (if female).
* Currently lactating and breast-feeding (if female).
* Inability to correctly answer all questions on the informed consent comprehension questionnaire.
* Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, or renal disease by history, physical examination, and/or laboratory studies.
* Behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the ability of the volunteer to understand and cooperate with the study protocol.
* Laboratory evidence of liver disease (alanine aminotransferase [ALT] greater than 64 U/l [females] or greater than 58 U/l [males]).
* Laboratory evidence of renal disease (serum creatinine greater than 1.1 mg/dl [females] or greater than 1.3 mg/dl [males], or more than trace protein or blood on urine dipstick testing).
* Laboratory evidence of hematologic disease (absolute leukocyte count <3000/mm3 or >12.5 x 103/mm3; hemoglobin <10.3 g/dl [females] or <11.0 g/dl [males]; absolute lymphocyte count <900/mm3; or platelet count <120,000/mm3).
* Other condition that in the opinion of the investigator would jeopardize the safety or rights of a volunteer participating in the trial or would render the subject unable to comply with the protocol.
* Participation in another investigational vaccine or drug trial within 30 days of starting this study.
* Volunteer has had medical, occupational, or family problems as a result of alcohol or illicit drug use during the past 12 months.
* History of a severe allergic reaction or anaphylaxis.
* Severe asthma as defined by the need for regular use of inhalers or emergency clinic visit or hospitalization within the last 6 months.
* Positive ELISA for HCV.
* Positive ELISA for HBsAg.
* Known immunodeficiency syndrome.
* Use of corticosteroids (excluding topical or nasal) or immunosuppressive drugs within 30 days of starting this study.
* Receipt of a live vaccine within past 4 weeks or a killed vaccine within past 2 weeks prior to entry into the study.
* History of a surgical splenectomy.
* Receipt of blood products within the past 6 months.
* Previous receipt of a primary series of any hepatitis B vaccine.
* History of allergy to yeast.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2007-05; Primary Completion 2008-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
To determine the frequency of vaccine-related adverse events, graded by severity, for each dose of the Na-ASP-2 Hookworm Vaccine | For the duration of the study

SECONDARY OUTCOMES:
To determine the dose of Na-ASP-2 that generates the highest antibody response as determined by an indirect enzyme-linked immunosorbent assay (ELISA) | 2 weeks after the third injection
To assess and compare the duration of antibody response to Na-ASP-2 | For the duration of the study
To perform exploratory studies of the cellular immune responses to the Na-ASP-2 antigen both before and after immunization | For the duration of the study

CONTACTS AND LOCATIONS:
Overall Officials: David J Diemert, MD, Principal Investigator — Albert B. Sabin Vaccine Institute
Locations (1):
- Centro de Pesquisas Rene Rachou, Belo Horizonte, Brazil

REFERENCES:
- [Result] Diemert DJ, Pinto AG, Freire J, Jariwala A, Santiago H, Hamilton RG, Periago MV, Loukas A, Tribolet L, Mulvenna J, Correa-Oliveira R, Hotez PJ, Bethony JM. Generalized urticaria induced by the Na-ASP-2 hookworm vaccine: implications for the development of vaccines against helminths. J Allergy Clin Immunol. 2012 Jul;130(1):169-76.e6. doi: 10.1016/j.jaci.2012.04.027. Epub 2012 May 26. PMID 22633322
- See also: Sponsor's Web page — http://www.sabin.org
- See also: Trial site website — http://www.cpqrr.fiocruz.br